CLINICAL TRIAL: NCT04253587
Title: Cognitive Intervention to Restore Capabilities for Learning and Retrieval of High-Fidelity Memory
Brief Title: Wayfinding Intervention in High-Fidelity Long-Term Memory
Acronym: LABYR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-27586-A
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Long-Term Memory Decline; Mild Cognitive Impairment
Keywords: amnestic MCI without dementia; cognitive training
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Tomography, Optical Coherence; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: After recruitment, participants are randomly assigned to treatment arms. Participants and experimenters with whom they interact during the experiments are blind to the purpose of the randomly-assigned arm. First-level analysis performed blind to participant's treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (6):
- LabyrinthVR Trackers (Experimental): Multi-session cognitive intervention with head-mounted display virtual reality computer game that presents an adaptive spatial wayfinding challenge. Game movement via participant ambulation wearing leg-position trackers.
  Interventions: Device: LabyrinthVR
- LabyrinthVR Scoot (Experimental): Multi-session cognitive intervention with head-mounted display virtual reality computer game that presents an adaptive spatial wayfinding challenge. Game movement via teleporting technique.
  Interventions: Device: LabyrinthVR
- Placebo Controls (Placebo Comparator): Multi-session cognitive intervention with handheld tablet or wireless virtual reality headset presentation of commercially available, narrative computer games.
  Interventions: Device: Placebo Games
- Coherence (Active Comparator): Multi-session cognitive intervention with head-mounted display virtual reality computer game that presents an adaptive rhythm training game.
  Interventions: Device: Coherence
- Labyrinth Tablet (Experimental): Multi-session cognitive intervention with tablet computer, displaying 2.5D version of Labyrinth game in an adaptive spatial wayfinding challenge. Game movement via on-screen control buttons.
  Interventions: Device: Tablet
- Labyrinth VR wireless (Experimental): Multi-session cognitive intervention with head-mounted display virtual reality computer game using wireless, narrower filed technology to presents an adaptive spatial wayfinding challenge. Game movement via teleporting technique.
  Interventions: Device: LabyrinthVR

INTERVENTIONS:
Device: LabyrinthVR — Head-mounted display virtual reality game designed to induce environmental enrichment in an adaptive, immersive regimen of wayfinding in novel urban and village neighborhoods.
  Arms: Labyrinth VR wireless; LabyrinthVR Scoot; LabyrinthVR Trackers
Device: Placebo Games — Commercially-available, narrative computer games marketed as cognitively enriching.
  Arms: Placebo Controls
Device: Coherence — Head-mounted display virtual reality game designed to present an adaptive rhythm training routine.
  Arms: Coherence
Device: Tablet — Tablet computer playing Labyrinth VR game but in 2.5D
  Arms: Labyrinth Tablet

SUMMARY:
Therapeutic treatment is yet available for declining memory, which is an impairment affecting the quality of life for many older adults and patients with cognitive impairment. Cognitive training with an immersive video game promises to drive hippocampal-cortical plasticity and associated gains that can restore memory capability or provide therapeutic treatment for memory deficits.

DETAILED DESCRIPTION:
A hallmark of higher cognition is the capability for flexible association of diverse bits of information stored in memory, such that experiences can be remembered in detailed and distinct terms (i.e., high-fidelity long-term memory (LTM)). Interventions capable of sustaining improved learning and flexible association of new information into LTM remain elusive. Interventions have yet to be developed to attenuate the decline of high-fidelity LTM in normal aging or provide therapeutic treatment for patients with cognitive impairment without dementia (i.e., MCI).

This project applies a translational neuroscience approach in development of a cognitive training intervention that targets sustained improvement in capabilities for LTM and cognitive control. Treatments use commercially available head-mounted display Virtual Reality (VR) technology and tablet computers to present a deeply immersive spatial wayfinding video game. Based on preliminary results, the hypothesis is that immersion in a game to navigate errands through unfamiliar, visually complex neighborhoods (i.e., wayfinding) will be an effective means to environmental enrichment, which refers to a process whereby new and complex experiences bring change to brain and behavior.

The significance of this platform is from the effects in brain and behavior arising from cognitive training, which can generalize to improvements in untrained capability for high-fidelity LTM. Research in rodents and humans shows that learning a new, enriched environment spurs the healthy function of the hippocampus and supports lifelong neurogenesis. Adult-borne hippocampal neurogenesis has been linked as the neurobiological basis for the formation of new, high-fidelity memories.

The Labyrinth spatial wayfinding game was developed in-house to incorporate full scientific rigor, as with procedures in any properly controlled behavioral experiment. The game uses 3D and 2.5D computer graphics tools, as well as numerous levels of adaptive challenge, to deliver a dynamic, engaging experience for participants throughout the training regimen. Training can be administered with and without participant ambulation in movement through wayfinding runs.

A participant's pre- and post-training assessments will occur promptly before and after their 15 to 20-hour training regimen, including collection of functional MRI (fMRI) and structural MRI data. Cognitive outcome measures will assess capabilities for high-fidelity LTM retrieval.

The a priori hypothesis is that effectiveness of the wayfinding game intervention would be evidenced by post-training improvements in retrieval of high-fidelity LTM and associated cognitive control capabilities. FMRI results associated with the measured cognitive improvements will localize changes in functional brain networks that support gains in memory capabilities. Structural MRI measures will assess morphometric and volumetric changes from pre- to post-training assessments.

ELIGIBILITY:
Inclusion Criteria:

* fluent speakers of English
* completed 12 or more years of education
* normal or corrected-to-normal vision
* dexterity to comfortably operate the scanner-compatible response box
* freedom from physical and neurological conditions contra-indicated for fMRI
* must confirm physical stamina and comfort for 45-minute, brisk walks on level ground

Exclusion Criteria:

* use of psychotropic medications
* history of concussions or dizziness, vestibular or balance problems
* significant discomfort with virtual reality experiences

Ages: 62 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Wais, PhD, Principal Investigator — Neuroscape, Department of Neurology
Locations (1):
- UCSF Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wais PE, Arioli M, Anguera-Singla R, Gazzaley A. Virtual reality video game improves high-fidelity memory in older adults. Sci Rep. 2021 Jan 28;11(1):2552. doi: 10.1038/s41598-021-82109-3. PMID 33510315

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LabyrinthVR Trackers | Placebo Controls
Started | 25 | 25
Baseline T1 | 24 | 21
Post Training T2 | 21 | 21
Completed | 21 | 21
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- LabyrinthVR Trackers: Participants who completed the intervention active training game using head-mounted display virtual reality headset.
- Placebo Controls: Participants who completed the intervention control games using a tablet computer.
- Total: Total of all reporting groups
Arm/Group | LabyrinthVR Trackers | Placebo Controls | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 23 | 20 | 43
Age, Continuous [Mean (Full Range); unit: years] — The key participant variable was age.
  years | 69.1 [64 to 81] | 68.3 [63 to 79] | 68.7 [63 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 16 | 12 | 28
  Unknown or Not Reported | 6 | 8 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: MDT Change in Mnemonic Discrimination
Description: Mnemonic discrimination task testing recognition memory for common objects, as reported in scores on a scale of the Lure Discrimination Index ranging from 0.00 to 1.00 where higher values show better performance.
Time Frame: baseline immediately before and post-assessment immediately after training regimen is completed
Measure: Mean (Standard Error); unit: LDI score on a scale
Arm/Group | LabyrinthVR Trackers | Placebo Controls
Number analyzed (Participants) | 21 | 21
LDI score on a scale | 0.09 (0.03) | 0.01 (0.03)
Statistical Analysis 1: Comparison: LabyrinthVR Trackers vs Placebo Controls; Test type: Equivalence — The null hypothesis was no difference between mean change scores for time-points X conditions; p = 0.016, ANOVA — Mixed effects ANOVA applied family wise error for post-hoc tests according to a priori hypothesis; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.06 to 0.06], Standard Error of Mean 0.03

2. Primary Outcome: WALK Change in Recall
Description: Encoding and test of recent autobiographical long-term memory, as reported in scores on a scale of Percentage of Items Recalled ranging from 0.00 to 1.00 where higher values show better performance.
Time Frame: baseline immediately before and post-assessment immediately after training regimen is completed
Measure: Mean (Standard Error); unit: Items Recalled score on a scale
Arm/Group | LabyrinthVR Trackers | Placebo Controls
Number analyzed (Participants) | 21 | 21
Items Recalled score on a scale | 0.03 (0.02) | 0.00 (0.02)
Statistical Analysis 1: Comparison: LabyrinthVR Trackers vs Placebo Controls; Test type: Superiority; p = 0.22, ANOVA; effect of condition (F1,20 = 1.616, p = 0.22), effect of time (F1,20 = 0.613, p = 0.44); Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.03 to 0.03], Standard Error of Mean 0.035

3. Primary Outcome: Changes in Volumetric-based Brain Morphometry Associated With Training-induced Changes in Mnemonic Discrimination
Description: Structural MRI T1 data will be analyzed in terms of volumetric-based morphometry and compared between treatment arms and timepoints.
Time Frame: during collection of Outcome 1, baseline immediately before and post-assessment immediately after training regimen is completed
Population: THESE DATA WERE NOT COLLECTED OR ANALYZED DUE TO FUNDING CONSTRAINTS
Arm/Group | LabyrinthVR Trackers | Placebo Controls
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Changes in Task-based Cortical Functional Connectivity Associated With Training-induced Changes in Mnemonic Discrimination
Description: functional MRI data will be analyzed in terms of beta-series correlations between co-active cortical regions of interest and compared between treatment arms and timepoints.
Time Frame: as for outcome 3
Population: THESE DATA WERE NOT COLLECTED OR ANALYZED DUE TO FUNDING CONSTRAINTS
Arm/Group | LabyrinthVR Trackers | Placebo Controls
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Remote Cognitive Module (RCM)
Description: A tablet application using a speech-to-text interface to administer neuropsychological tests comparable to CVLT-II verbal memory, verbal fluency, digit span and Trail Making Test-B.
  Raw scores from the tasks will be transformed to z-scores, relative to population normative values, and a participant's z-scores will be the uniform measures of their performance across RCM tasks.
  THESE DATA WERE NOT COLLECTED OR ANALYZED DUE TO FUNDING CONSTRAINTS
Time Frame: baseline immediately before and post-assessment immediately after training regimen is completed
Population: THESE DATA WERE NOT COLLECTED OR ANALYZED DUE TO FUNDING CONSTRAINTS
Arm/Group | LabyrinthVR Trackers | Placebo Controls
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Test of Visual Attention Change in Top-down Control
Description: test of speed and accuracy of visual attention and impulsivity
Time Frame: baseline immediately before and post-assessment immediately after training regimen is completed
Population: THESE DATA WERE NOT COLLECTED OR ANALYZED DUE TO FUNDING CONSTRAINTS
Arm/Group | LabyrinthVR Trackers | Placebo Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Over the total study period of 18 months, individual participants were observed during an approximate six-week period from baseline through post-training assessments.
Arm/Group | LabyrinthVR Trackers | Placebo Controls
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT04253587/Prot_SAP_001.pdf